CLINICAL TRIAL: NCT05118360
Title: A Seamless Phase 2a/2b, Double-Blind, Randomized, Multicenter, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of ASC41, a Thyroid Hormone Receptor β Agonist, in Adults With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of ASC41 in Adults With NASH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been cancelled due to business reasons
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC41-201
Record Dates: First submitted 2021-11-01; First posted 2021-11-12 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: NAFLD; Phase 2; Thyroid hormone receptor agonist; NASH; ASC41
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Randomized in 2:1 ratio to receive either oral ASC41 2 mg or oral matching placebo. Randomized in 2:1 ratio to receive either oral ASC41 4 mg or oral matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1-ASC41 2mg (Experimental): ASC41 2mg for 52 weeks.
  Interventions: Drug: ASC41 2 mg
- Part1-placebo (Placebo Comparator): Matching placebo for 52 weeks.
  Interventions: Drug: Placebo
- Part 2-ASC41 4mg (Experimental): ASC41 4 mg for 52 weeks.
  Interventions: Drug: ASC41 4 mg
- Part2-placebo (Placebo Comparator): Matching placebo for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC41 2 mg — 2mg of ASC41 orally once daily for 52 weeks
  Arms: Part 1-ASC41 2mg
Drug: ASC41 4 mg — 4mg of ASC41 orally once daily for 52 weeks
  Arms: Part 2-ASC41 4mg
Drug: Placebo — Matching placebo orally once daily for 52 weeks.
  Arms: Part1-placebo; Part2-placebo

SUMMARY:
This is a phase 2, randomized, double-blind, placebo controlled study in adults with biopsy confirmed NASH. The study is aimed at evaluating efficacy and tolerability of ASC41 in adults with NASH.

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of ≥ 8% liver fat content on screening MRI-PDFF.
* Histologic evidence of NASH upon central read of a liver biopsy obtained no more than 6 months before Day 1 defined by NASH activity score (NAS) greater than or equal to 4 with at least 1 point each in inflammation and ballooning.
* Diabetes Mellitus well controlled based on laboratory test HbA1c ≤ 9.5%.

Key Exclusion Criteria:

* Evidence of advanced liver disease such as cirrhosis (stage 4 fibrosis) or decompensated liver disease (e.g. ascites, esophageal varices) or liver cancer.
* Evidence of other causes of chronic liver disease.
* Weight change ≥ 5% after qualifying liver biopsy or MRI-PDFF performed.
* Any contraindications to a MRI scan.
* Treatment with vitamin E (unless stable dose of < 400 IU/d), thiazolidinediones (TZD), or glucagon-like peptide-1 receptor agonists (GLP-1 RA), unless subject is on a stable dose for 6 months prior to qualifying liver biopsy.
* Known history of alcohol or other substance abuse within the last year or at any time during the study.
* Use of any investigational drug within 6 months of MRI-PDFF and/or liver biopsy.
* Known positivity for antibody to Human Immunodeficiency Virus (HIV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-10 (Estimated); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Percent of ASC41 subjects compared to placebo with histological reduction in NAS ≥2 points that results from reduction of inflammation or ballooning and no worsening fibrosis assessed by histopathological reading of liver biopsy at Week 52 | Baseline to Week 52

SECONDARY OUTCOMES:
Safety and tolerability of ASC41 evaluated by incidence of treatment emergent adverse events (TEAEs) in ASC41 treated subjects compared to placebo | Baseline to Week 52
Change in hepatic fat fraction based on MRI-PDFF measurements in ASC41 treated subjects compared to placebo. | Baseline to Week 12 and Week 52
Resolution of NASH on overall histopathological reading of liver biopsy specimen taken at Week 52 compared to baseline in ASC41 treated subjects compared to placebo treated subjects | Baseline to Week 52